CLINICAL TRIAL: NCT06067932
Title: Mid- and Forefoot Disorders in Adolescents and Adults With X-linked Hypophosphatemia
Brief Title: Foot Disorders in X-linked Hypophosphatemia
Status: Completed | Type: Observational
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Principal Investigator, Forian Wenzel-Schwarz, Orthopedic surgeon, Orthopedic Hospital Vienna Speising
Other Study IDs: Midfoot XLH
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: X-linked Hypophosphatemia
Keywords: foot and ankle
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Foot X rays — Radiographs of ankle and foot anteroposterior/dorsoplantar were taken in standing position with a centralized beam on the ankle joint.
Diagnostic Test: Clinical examination + scores — The American Orthopedic Foot and Ankle Society Score (AOFAS- midfoot section and 1st Forefoot ray, Forefoot ray 2-5) and the foot function index (FFI) were assessed

SUMMARY:
This study aimed to characterize foot pathologies using X-rays and clinical examination and assess related outcome scores in adolescents and adults with X-linked Hypophophatemia

DETAILED DESCRIPTION:
A single center, cross-sectional analysis of adolescent and adult patients with XLH with and without previous surgical intervention was performed at the Orthopaedic Hospital Speising, Vienna, Austria. Clinical examination, quality of life questionnaires and radiographic data of foot x-rays in standing position were collected. Radiographic evaluation was performed to analyze foot deformity as well as signs of osteoarthritis at the foot.

ELIGIBILITY:
Inclusion Criteria: - Patients with confirmed XLH, ≥ 16 years were invited to participate in this study

Exclusion Criteria:

* Exclusion criteria were other forms of hypophosphatemia, pregnancy and recent lower limb surgery within 3 months.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rare bone disease (XLH) with and without foot problems
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Number of feet with signs of osteoarthritis | baseline
  radiographic signs of osteoarthritis at the foot joints

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mindler, Dr, Study Chair — Orthopedic Hospital Speising Vienna
Locations (1):
- Orthopedic Hospital Speising Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No